CLINICAL TRIAL: NCT00002733
Title: ALPHA INTERFERON, TUMOR INFILTRATING LYMPHOCYTES, AND INTERLEUKIN-2 IN THE TREATMENT OF CANCER
Brief Title: Biological Therapy in Treating Patients With Metastatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Purpose: Treatment
Other Study IDs: CDR0000064631; CBRG-9510; NBSG-9510; NCI-V96-0835
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Kidney Cancer; Melanoma (Skin); Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV renal cell cancer; stage IV melanoma; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha; Cimetidine

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Biological: therapeutic tumor infiltrating lymphocytes
Drug: cimetidine

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining different types of biological therapies, including interferon alfa, interleukin-2, and tumor infiltrating lymphocytes, may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of biological therapies, including interferon alfa, interleukin-2, and tumor infiltrating lymphocytes, in treating patients with metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and failure-free survival in patients with metastatic cancer (preferably melanoma or renal cell) treated with autologous tumor infiltrating lymphocytes (TIL), interferon alfa (IFN-A), and interleukin-2 (IL-2). II. Describe the toxic effects and costs associated with this therapy to assess risk benefit and cost benefit. III. Assess the relative value of administering low- or high-dose TIL, as well as the value of administering IFN-A before TIL, IL-2 with TIL, or cimetidine with TIL.

OUTLINE: This is a multicenter study. Patients are stratified according to center, tumor infiltrating lymphocyte (TIL) dose (low vs high), and medical condition suitable for interferon alfa (IFN-A)/interleukin-2 (IL-2) (yes vs no). Patients are assigned to one of two treatment regimens based on entry criteria. Regimen A (preferred): Patients meeting the preferred entry criteria receive IFN-A subcutaneously on days 1-4, TIL expanded in vitro with IL-2 IV on day 5, and IL-2 IV continuously over 72 hours following TIL infusion. Regimen B: All other patients receive TIL infusion once followed by oral cimetidine every 6 hours for 4 weeks. Treatment repeats in both regimens every 3-6 weeks in the absence of disease progression and according to TIL availability. Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 20-30 patients with melanoma and 20-30 patients with renal cell carcinoma will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologic evidence of any type of cancer with metastases Melanoma or renal cell cancer preferred No active brain metastasis Tumor infiltrating lymphocytes must be available Measurable or evaluable disease preferred

PATIENT CHARACTERISTICS: Age: 18 and over (under 75 preferred) Performance status: ECOG 0-3 (ECOG 0 or 1 preferred) Hematopoietic: (preferred) WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hematocrit at least 30% (transfusion allowed) Hepatic: (preferred) Bilirubin less than 2.0 mg/dL PT/PTT normal Renal: (preferred) Creatinine less than 2.0 mg/dL Cardiovascular: (preferred) At least 6 months since prior myocardial infarction No congestive heart failure, cardiac arrhythmia, or hypertension requiring medication Pulmonary: (preferred) pO2 at least 60 mm Hg Reasonable respiratory reserve No supplemental oxygen requirement Not dyspneic at rest Other: No chronic auto-coagulation (preferred) No active infection No chronic underlying immunodeficiency disease (including HIV, hepatitis B) No known autoimmune disease Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy (7 days since stereotactic radiosurgery) Surgery: At least 4 weeks since prior surgery to control brain metastases No prior organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1996-01; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

REFERENCES:
- [Background] Dillman RO, Hurwitz SR, Schiltz PM, Barth NM, Beutel LD, Nayak SK, O'Connor AA. Tumor localization by tumor infiltrating lymphocytes labeled with indium-111 in patients with metastatic renal cell carcinoma, melanoma, and colorectal cancer. Cancer Biother Radiopharm. 1997 Apr;12(2):65-71. doi: 10.1089/cbr.1997.12.65. PMID 10851449
- [Background] Schiltz PM, Beutel LD, Nayak SK, Dillman RO. Characterization of tumor-infiltrating lymphocytes derived from human tumors for use as adoptive immunotherapy of cancer. J Immunother. 1997 Sep;20(5):377-86. doi: 10.1097/00002371-199709000-00007. PMID 9336745
- [Background] Dillman RO, Hurwitz R, Schlitz PM, et al.: Radioimmunodetection of cancer with 111-Indium conjugated tumor infiltrating lymphocytes in patients with metastatic renal cell carcinoma. J Immunother 19(6): 457, 1996.